CLINICAL TRIAL: NCT06892704
Title: Olfactory Cleft Obstruction and Electrophysiological Olfactory Bulb Generated Beta Field Potentials Predict Olfactory Restoration by Dupilumab in CRSwNP Patients.
Brief Title: Olfactory Cleft Obstruction and Electrophysiological Field Potentials Predict Olfactory Restoration by Dupilumab in CRSwNP Patients.
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: STU0022296
Record Dates: First submitted 2025-03-19; First posted 2025-03-25 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Chronic Rhinosinusitis Phenotype With Nasal Polyps (CRSwNP); Smell Loss
Keywords: Dupilumab; Chronic Rhinosinusitis with Nasal Polyps; Smell Loss; Electrophysiology
MeSH Terms: conditions — Anosmia | interventions — dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Nasal secretions, Exhaled Breath Condensate, Tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Dupilumab Treatment: Patients who had prior endoscopic sinus surgery for CRSwNP with persistent smell loss initiating dupilumab
  Interventions: Drug: Dupilumab - Standard Dose

INTERVENTIONS:
Drug: Dupilumab - Standard Dose — 24 weeks of dupilumab 300mg q2 weeks

SUMMARY:
The goal of this observational study is to learn what can predict the return of the sense of smell in patients with chronic rhinosinusitis with nasal polyps being treated with dupilumab. The main questions it aims to answer are:

1. Does obstruction of the olfactory cleft predict return of the sense of smell?
2. Do electrophysiological signals generated by breathing and sniffing behavior predict return of the sense of smell?

Participants starting dupilumab will undergo assessment for their degree of olfactory cleft obstruction, and an electrophysiologic assessment of their olfactory cleft and be followed over 6 months of treatment with dupilumab.

ELIGIBILITY:
* Well documented history of CRSwNP
* BSIT age/sex classified as "abnormal" score
* Self-reported stable olfactory deficit of moderate to severe quality > 3 months
* Prior endoscopic sinus surgery >3 months, <10 years prior

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a well documented history of CRSwNP who had prior endoscopic sinus surgery who experience and are assessed to have olfactory deficit.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Status change of the Brief Smell Identification Test | 26 weeks
  The brief smell identification test will be administered and patients classified into normal/age-related deficit vs abnormal.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University Feinberg School of Medicine, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD underlying publication
Supporting Information: Study Protocol